CLINICAL TRIAL: NCT02500979
Title: A Randomized, Single-Blind, Two-Way Crossover, Placebo-Controlled Phase I Study to Compare the 24-hour Glucose Profile and Safety of Pramlintide and Insulin, Co-Administered in a Fixed-Dose Ratio, Versus Placebo and Insulin in Patients With Type 1 Diabetes Mellitus With Inadequate Glycemic Control
Brief Title: Effect of a Fixed Pramlintide: Insulin Dose Ratio on Postprandial Glucose in Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: D5570C00002
Record Dates: First submitted 2015-07-10; First posted 2015-07-17 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-03

CONDITIONS: Type 1 Diabetes Mellitus
Keywords: Type 1 Diabetes Mellitus; Pramlintide
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — pramlintide; Insulin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pramlintide acetate & regular insulin (Experimental): Pramlintide will be adiministered by sc infusion at a concentration of 1000ug/mL
  Interventions: Drug: Pramlintide acetate; Drug: Lispro insulin U-100; Drug: Regular insulin U-100
- Placebo and regular insulin (Placebo Comparator): Placebo is similar sterile solution without pramlintide.
  Interventions: Drug: Placebo; Drug: Lispro insulin U-100; Drug: Regular insulin U-100

INTERVENTIONS:
Drug: Pramlintide acetate — Pramlintide acetate administered by a separate pump
  Other Names: Pramlintide: SYMLIN
  Arms: Pramlintide acetate & regular insulin
Drug: Placebo — Placebo administered by separate pump
  Arms: Placebo and regular insulin
Drug: Lispro insulin U-100 — Subjects will be stabilized on a separate insulin pump and administered lispro insulin throughout the study, except during both inpatient treatment periods (Visit 4 and Visit 5)
  Other Names: Humalog insulin lispro U-100
Drug: Regular insulin U-100 — Use during two in-patient treatment periods (visits 4 and 5) and administered by separate pump
  Other Names: Humulin R; U-100

SUMMARY:
This study is designed to investigate the clinical efficacy and safety of pramlintide co-administered as a fixed-dose ratio with basal-bolus SC insulin, delivered simultaneously via 2 separate pumps, in subjects with type 1 diabetes who are failing to achieve the desired level of glycemic control using insulin therapy.

DETAILED DESCRIPTION:
Potentially eligible subjects with Type 1 diabetes mellitus who are treated with with a basal-bolus insulin regimen through multiple daily injections or insulin pump at a total daily insulin dose ≤60 U, will be eligible. Visit 1 is approximately 3-6 weeks prior to randomization. Given some variability in HbA1c and C-peptide assays, re-testing for HbA1c and C-peptide can be performed within 18 days from the initial visit. Visit 2 is approximately 2-5 weeks prior to randomization. Subjects are on lispro insulin throughout study except during Visit 4 and Visit 5, the domicile 24 hr treatment period, when they are switched to regular insulin U-100.

Screen failed patients may be re-screened for inclusion in the study, as long as re-screening takes place at least 3 months after the original screening visit. If a subject is re-screened, he/she must continue to meet all inclusion/exclusion criteria. All study procedures of initial Visit 1 must be repeated at the re-screening visit.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study-specific procedures
* Female and/or male aged between 18 and 70 years
* Must have a prior diagnosis of T1DM
* Body mass index (BMI) <30 kg/m2
* Subjects are not on current treatment with pramlintide (Symlin) and have not received pramlintide during the 6-month period prior to enrollment
* Subjects should be willing to consume all of the components of the standardized meals administered during the study
* Negative serum pregnancy test for female subjects of childbearing potential
* Female subjects of childbearing potential must be 1 year postmenopausal, surgically sterile, or using an acceptable method of contraception for the duration of the study
* Male subjects must be surgically sterile or using an acceptable method of contraception for the duration of the study

Exclusion Criteria:

* Recurrent severe hypoglycemia requiring assistance within 6 months before screening
* A history of hypoglycemia unawareness
* A confirmed diagnosis of gastroparesis
* Has been treated, is currently being treated, or is expected to require or undergo treatment with the following medications:
* Any oral antihyperglycemic agent or any other injectable antihyperglycemic agent that is not insulin
* Drugs that directly affect GI motility (eg, anticholinergic agents such as atropine)
* Drugs that slow the intestinal absorption of nutrients (eg, α-glucosidase inhibitors
* A history of gastric surgery (such as gastric banding, Roux- and Y bypass)
* Is expected to require or undergo treatment with acetaminophen after enrollment and at any point during the study
* Has experienced diabetic ketoacidosis within the last 24 weeks
* History of hospitalization within the last 6 months for glycemic control (for both hyperglycemia or hypoglycemia)
* Subject has any significant disease or disorder, which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or may influence the results of the study, or the subject's ability to participate in the study
* Any clinically relevant abnormal findings, which, in the opinion of the investigator, may put the subject at risk because of his/her participation in the study.
* Pregnancy confirmed by a positive pregnancy test, or otherwise verified.
* Breast feeding
* Positive hepatitis C virus antibody (HCV Ab), hepatitis B virus surface antigen (HBsAg), hepatitis B virus core antibody (anti-Hbc), or human immunodeficiency virus 1/2 antibody (HIV-1/2 Ab) at Screening
* History of, or current alcohol or drug abuse
* Has donated blood within 2 months of Visit 1 (Screening) or is planning to donate blood during the study
* Has had a major surgery or a blood transfusion within 2 months before Visit 1 (screening)
* Participation in any clinical study with an investigational drug or new formulation of a marketed drug during the last 1 month prior to Visit 1

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2015-08-17 (Actual); Primary Completion 2016-08-05 (Actual); Study Completion 2016-08-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter Ohman, MD, Study Director — Medical Director AstraZeneca
Locations (3):
- United States (3):
  - Research Site, Chula Vista, California
  - Research Site, Portland, Oregon
  - Research Site, Chattanooga, Tennessee

REFERENCES:
- [Derived] Riddle MC, Nahra R, Han J, Castle J, Hanavan K, Hompesch M, Huffman D, Strange P, Ohman P. Control of Postprandial Hyperglycemia in Type 1 Diabetes by 24-Hour Fixed-Dose Coadministration of Pramlintide and Regular Human Insulin: A Randomized, Two-Way Crossover Study. Diabetes Care. 2018 Nov;41(11):2346-2352. doi: 10.2337/dc18-1091. Epub 2018 Sep 13. PMID 30213882

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The first subject was enrolled in the study (at Visit 2) on 27 August 2015. A total of 79 subjects were screened and 34 subjects were randomized at 3 sites in the United States. One additional subject was randomized in error and was discontinued prior to receiving any study medication. The last subject completed the study on 05 August 2016.
Pre-assignment Details: Eligible study subjects were males and females, aged ≥18 years and ≤70 years at the time of screening with a prior diagnosis of type 1 diabetes mellitus (T1DM) and an HbA1c value of ≥7.2% and ≤9.0% at screening.
Groups:
- Pramlintide First, Then Placebo: (Treatment Sequence A)
- Placebo First, Then Pramlintide: (Treatment Sequence B)
Period: Period 1
Arm/Group | Pramlintide First, Then Placebo | Placebo First, Then Pramlintide
Started ((Randomized Analysis Set)) | 16 | 17
Completed (Number of subjects that entered Period 2) | 12 | 16
Not Completed | 4 | 1
Not completed — Hyperglycemia | 1 | 0
Not completed — Severe non-compliance to protocol | 0 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Subject decision | 2 | 0
Period: Period 2
Arm/Group | Pramlintide First, Then Placebo | Placebo First, Then Pramlintide
Started ((Randomized Analysis Set)) | 12 | 16
Completed (Completed Period 2) | 11 | 16
Not Completed | 1 | 0
Not completed — Change in risk | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All randomized subjects receiving any infused study treatment. Subjects were analyzed according to the treatment sequence they received.
Groups:
- Pramlintide First, Then Placebo: (Treatment Sequence A) - Safety Analysis Set
- Placebo First, Then Pramlintide: (Treatment Sequence B) - Safety Analysis Set
- Total: Total of all reporting groups
Arm/Group | Pramlintide First, Then Placebo | Placebo First, Then Pramlintide | Total
Number analyzed (Participants) | 16 | 16 | 32
Age, Categorical [Count of Participants; unit: Participants] — Population: Safety Analysis Set: All randomized subjects receiving any infused study treatment. Subjects were analyzed according to the treatment sequence they received.
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 14 | 16 | 30
    >=65 years | 2 | 0 | 2
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Safety Analysis Set: All randomized subjects receiving any infused study treatment. Subjects were analyzed according to the treatment sequence they received.
  Years | 45.1 (14.83) | 38.9 (12.68) | 42.0 (13.92)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Safety Analysis Set: All randomized subjects receiving any infused study treatment. Subjects were analyzed according to the treatment sequence they received.
  Participants
    Female | 13 | 12 | 25
    Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Safety Analysis Set: All randomized subjects receiving any infused study treatment. Subjects were analyzed according to the treatment sequence they received.
  Participants
    Hispanic or Latino | 0 | 2 | 2
    Not Hispanic or Latino | 16 | 14 | 30
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Safety Analysis Set: All randomized subjects receiving any infused study treatment. Subjects were analyzed according to the treatment sequence they received.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 0 | 1
    White | 15 | 15 | 30
    More than one race | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kg] — Population: Safety Analysis Set: All randomized subjects receiving any infused study treatment. Subjects were analyzed according to the treatment sequence they received.
  kg | 72.03 (9.012) | 68.73 (8.859) | 70.38 (8.949)
Height [Mean (Standard Deviation); unit: cm] — Population: Safety Analysis Set: All randomized subjects receiving any infused study treatment. Subjects were analyzed according to the treatment sequence they received.
  cm | 168.41 (6.966) | 167.31 (7.684) | 167.86 (7.236)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] — Population: Safety Analysis Set: All randomized subjects receiving any infused study treatment. Subjects were analyzed according to the treatment sequence they received.
  kg/m^2 | 25.38 (2.806) | 24.52 (2.341) | 24.95 (2.579)
Duration of Diabetes [Mean (Standard Deviation); unit: Years] — Population: Safety Analysis Set: All randomized subjects receiving any infused study treatment. Subjects were analyzed according to the treatment sequence they received.
  Years | 27.81 (13.177) | 21.94 (10.866) | 24.88 (12.249)
Current Administration of Insulin [Count of Participants; unit: Participants] — Subject's usual method of insulin administration - either multiple daily injections (MDI) or continuous subcutaneous infusion of insulin (CSII), or both. Population: Safety Analysis Set: All randomized subjects receiving any infused study treatment. Subjects were analyzed according to the treatment sequence they received.
  Participants
    CSII | 10 | 11 | 21
    MDI | 4 | 5 | 9
    Both | 2 | 0 | 2
Renal Status Category [Count of Participants; unit: Participants] — Population: Safety Analysis Set: All randomized subjects receiving any infused study treatment. Subjects were analyzed according to the treatment sequence they received.
  Participants
    <30 mL/min | 0 | 0 | 0
    ≥30 to <60 mL/min | 2 | 0 | 2
    ≥60 to <90 mL/min | 8 | 8 | 16
    ≥90 mL/min | 6 | 8 | 14
Baseline Fasting Glucose [Mean (Standard Deviation); unit: mmol/L] — Population: Safety Analysis Set: All randomized subjects receiving any infused study treatment. Subjects were analyzed according to the treatment sequence they received.
  mmol/L
    number analyzed (Participants) | 15 | 16 | 31
    (all) | 8.57 (2.767) | 8.15 (3.149) | 8.35 (2.928)
Baseline A1c [Mean (Standard Deviation); unit: %] — Population: Safety Analysis Set: All randomized subjects receiving any infused study treatment. Subjects were analyzed according to the treatment sequence they received.
  % | 7.84 (0.356) | 8.21 (0.574) | 8.03 (0.506)
Baseline C-peptide [Mean (Standard Deviation); unit: nmol/L] — Population: Safety Analysis Set: All randomized subjects receiving any infused study treatment. Subjects were analyzed according to the treatment sequence they received.
  nmol/L
    number analyzed (Participants) | 1 | 2 | 3
    (all) | 0.030 (0) | 0.030 (0.0141) | 0.030 (0.0100)
Baseline Insulin [Mean (Standard Deviation); unit: U/day] — Population: Safety Analysis Set: All randomized subjects receiving any infused study treatment. Subjects were analyzed according to the treatment sequence they received.
  U/day | 38.14 (12.525) | 36.58 (8.920) | 37.36 (10.725)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Pramlintide by Measurement of 24-hour Tissue Mean Weighted Glucose (MWG) Obtained With Continuous Glucose Monitoring (CGM)
Description: 24-hour MWG mg/dL, defined as total area under the 24-hour tissue glucose curve obtained with CGM, divided by actual time span in the 24-hour period.
Time Frame: 24 h
Population: Full Analysis Set: Of the 33 correctly randomized subjects, 26 (76.5%) had at least 1 efficacy assessment available from each of the 2 crossover periods and were included in the Full Analysis Set.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Groups:
- Placebo & Regular Insulin: Placebo was similar sterile solution without pramlintide
- Pramlintide & Regular Insulin: Pramlintide was administered by sc infusion at a concentration of 1000ug/ml
Arm/Group | Placebo & Regular Insulin | Pramlintide & Regular Insulin
Number analyzed (Participants) | 26 | 26
mg/dL | 173.8 (8.17) | 152.2 (8.17)
Statistical Analysis 1: Comparison: Placebo & Regular Insulin vs Pramlintide & Regular Insulin; Test type: Superiority or Other; p = 0.0118, Linear mixed-effects model; Least squares mean difference = -21.5, 95% CI 2-sided [-37.8 to -5.2], Standard Error of Mean 7.88

2. Secondary Outcome: Efficacy of Pramlintide by Measurement of Absolute Plasma Glucose Area Under the Plasma Concentration-time Curve (AUC) Following Lunch
Description: Absolute postprandial plasma glucose AUC was measured for the first 3 hours (AUC0-3h) following lunch based on sample availability. (Sample times: 20 hours [lunch], 20 hours 45 min, 21 hours, 23 hours, 24 hours).
Time Frame: 3 hours
Population: Pharmacokinetic/Pharmacodynamic (PK/PD) Analysis Set: Of the 33 correctly randomized subjects, 26 (76.5%) subjects received at least 1 dose of pramlintide and had evaluable PD data and were, therefore, included in the PK/PD Analysis Set.
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L*h
Arm/Group | Placebo & Regular Insulin | Pramlintide & Regular Insulin
Number analyzed (Participants) | 25 | 24
mmol/L*h | 36.233 [31.427 to 41.039] | 28.336 [23.487 to 33.185]
Statistical Analysis 1: Comparison: Placebo & Regular Insulin vs Pramlintide & Regular Insulin; Test type: Superiority or Other; p = 0.0013, Linear mixed effects model; LS mean difference (pramlintide-placebo) = -7.897, 95% CI 2-sided [-12.356 to -3.438]

3. Secondary Outcome: Efficacy of Pramlintide by Measurement of Absolute Plasma Glucose Area Under the Plasma Concentration-time Curve (AUC) Following Dinner
Description: Absolute postprandial plasma glucose AUC (AUC0-2h) was measured for the first 2 hours following dinner based on sample availability. (Sample times: 2 hours [dinner], 2 hours 45 min, 3 hours, 4 hours).
Time Frame: 2 hours
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L*h
Arm/Group | Placebo & Regular Insulin | Pramlintide & Regular Insulin
Number analyzed (Participants) | 25 | 26
mmol/L*h | 23.247 [20.472 to 26.021] | 17.970 [15.231 to 20.709]
Statistical Analysis 1: Comparison: Placebo & Regular Insulin vs Pramlintide & Regular Insulin; Test type: Superiority or Other; p = 0.0091, Linear mixed effects model; LS mean difference (pramlintide-placebo) = -5.277, 95% CI 2-sided [-9.175 to -1.378]

4. Secondary Outcome: Efficacy of Pramlintide by Measurement of Absolute Plasma Glucose Area Under the Plasma Concentration-time Curve (AUC) Following Breakfast
Description: Absolute postprandial plasma glucose AUC (AUC0-2h) was measured for the first 2 hours following breakfast based on sample availability. (Sample times: 16 hours [breakfast], 16 hours 45 min, 17 hours, 18 hours).
Time Frame: 2 hours
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L*h
Arm/Group | Placebo & Regular Insulin | Pramlintide & Regular Insulin
Number analyzed (Participants) | 26 | 24
mmol/L*h | 23.535 [20.817 to 26.253] | 19.101 [16.280 to 21.922]
Statistical Analysis 1: Comparison: Placebo & Regular Insulin vs Pramlintide & Regular Insulin; Test type: Superiority or Other; p = 0.0057, Linear mixed effects model; LS mean difference (pramlintide-placebo) = -4.435, 95% CI 2-sided [-7.445 to -1.424]

5. Secondary Outcome: Efficacy of Pramlintide by Measurement of Incremental 24-hour Tissue Glucose Area Under the Plasma Concentration-time Curve (AUC) Obtained With Continuous Glucose Monitoring (CGM)
Description: Incremental (i.e., baseline-corrected) area under the 24-hour tissue glucose concentration curve (AUC0-24h) measured by continuous glucose monitoring (CGM) with a pre-test, non-fasting tissue glucose value as baseline. (Sample times: 0, 30 min, 2 hours [dinner], 2 hours 45 min, 3 hours, 4 hours, 9 hours, 12 hours, 14 hours, 16 hours [breakfast], 16 hours 45 min, 17 hours, 18 hours, 20 hours [lunch], 20 hours 45 min, 21 hours, 23 hours, 24 hours).
Time Frame: 24 h
Population: Full Analysis Set: Of the 33 correctly randomized subjects, 26 (76.5%) had at least 1 efficacy assessment available from each of the 2 crossover periods and were included in the Full Analysis Set,
Measure: Least Squares Mean (Standard Error); unit: mg/dL*min
Arm/Group | Placebo & Regular Insulin | Pramlintide & Regular Insulin
Number analyzed (Participants) | 26 | 26
mg/dL*min | 26243 (3379.8) | -2489 (3379.8)
Statistical Analysis 1: Comparison: Placebo & Regular Insulin vs Pramlintide & Regular Insulin; Test type: Superiority or Other; p < 0.0001, Linear mixed-effects model; Least squares mean difference = -28733, 95% CI 2-sided [-37326 to -20139], Standard Error of Mean 4163.6

6. Secondary Outcome: Efficacy of Pramlintide by Measurement of Absolute 24-hour Plasma Glucose Area Under the Plasma Concentration-time Curve (AUC)
Description: Absolute mean area under the 24-hour plasma glucose concentration curve, measured as total area under the curve (0 to 24 hours). (Sample times: 0, 30 min, 2 hours [dinner], 2 hours 45 min, 3 hours, 4 hours, 9 hours, 12 hours, 14 hours, 16 hours [breakfast], 16 hours 45 min, 17 hours, 18 hours, 20 hours [lunch], 20 hours 45 min, 21 hours, 23 hours, 24 hours).
Time Frame: 24 h
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L*h
Arm/Group | Placebo & Regular Insulin | Pramlintide & Regular Insulin
Number analyzed (Participants) | 26 | 26
mmol/L*h | 243.835 [220.032 to 267.638] | 215.417 [191.614 to 239.220]
Statistical Analysis 1: Comparison: Placebo & Regular Insulin vs Pramlintide & Regular Insulin; Test type: Superiority or Other; p = 0.0258, Linear mixed-effects model; LS mean difference = -28.418, 95% CI 2-sided [-53.099 to -3.737]

7. Secondary Outcome: Efficacy of Pramlintide by Measurement of Incremental 24-hour Plasma Glucose Area Under the Plasma Concentration-time Curve (AUC)
Description: Incremental (i.e., baseline-corrected) mean area under the 24-hour plasma glucose concentration curve, measured as total area under the curve (0 to 24 hours). (Sample times: 0, 30 min, 2 hours [dinner], 2 hours 45 min, 3 hours, 4 hours, 9 hours, 12 hours, 14 hours, 16 hours [breakfast], 16 hours 45 min, 17 hours, 18 hours, 20 hours [lunch], 20 hours 45 min, 21 hours, 23 hours, 24 hours).
Time Frame: 24 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mmol/L*h
Arm/Group | Placebo & Regular Insulin | Pramlintide & Regular Insulin
Number analyzed (Participants) | 26 | 26
mmol/L*h | 11.181 (67.6648) | -12.753 (70.0174)

8. Secondary Outcome: Efficacy of Pramlintide Measured by Percent Time Spent in the Range of >70 mg/dL to <180 mg/dL Tissue Glucose Obtained With Continuous Glucose Monitoring (CGM)
Description: Percent time spent in the normoglycemic range of tissue glucose concentrations between >70 mg/dL and <180 mg/dL, measured by CGM. (Sample times: 0, 30 min, 2 hours [dinner], 2 hours 45 min, 3 hours, 4 hours, 9 hours, 12 hours, 14 hours, 16 hours [breakfast], 16 hours 45 min, 17 hours, 18 hours, 20 hours [lunch], 20 hours 45 min, 21 hours, 23 hours, 24 hours).
Time Frame: 24 h
Population: Full Analysis Set:Of the 33 correctly randomized subjects, 26 (76.5%) had at least 1 efficacy assessment available from each of the 2 crossover periods and were included in the Full Analysis Set.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of time
Arm/Group | Placebo & Regular Insulin | Pramlintide & Regular Insulin
Number analyzed (Participants) | 26 | 26
Percentage of time | 43.8 [33.6 to 56.9] | 57.2 [44.0 to 74.4]
Statistical Analysis 1: Comparison: Placebo & Regular Insulin vs Pramlintide & Regular Insulin; Test type: Superiority or Other; p = 0.0456, Linear mixed-effects model; LS Mean Ratio (Pramlintide/Placebo) = 1.31, 95% CI 2-sided [1.01 to 1.70]

9. Secondary Outcome: Efficacy of Pramlintide by Measurement of Absolute 24-hour Plasma Glucagon Area Under the Plasma Concentration-time Curve (AUC)
Description: Absolute mean area under the 24-hour plasma glucagon concentration curve, measured as total area under the curve (total AUC0-24). (Sample times: 0, 30 min, 2 hours [dinner], 2 hours 45 min, 3 hours, 4 hours, 9 hours, 12 hours, 14 hours, 16 hours [breakfast], 16 hours 45 min, 17 hours, 18 hours, 20 hours [lunch], 20 hours 45 min, 21 hours, 23 hours, 24 hours).
Time Frame: 24 h
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: h*pmol/L
Arm/Group | Placebo & Regular Insulin | Pramlintide & Regular Insulin
Number analyzed (Participants) | 26 | 26
h*pmol/L | 506.265 [459.096 to 558.280] | 481.633 [436.759 to 531.118]
Statistical Analysis 1: Comparison: Placebo & Regular Insulin vs Pramlintide & Regular Insulin; Test type: Superiority or Other; p = 0.1015, Linear mixed-effects model; LS mean ratio (pramlintide/placebo) = 0.951, 95% CI 2-sided [0.896 to 1.011]

10. Secondary Outcome: Efficacy of Pramlintide by Measurement of Incremental 24-hour Plasma Glucagon Area Under the Plasma Concentration-time Curve (AUC)
Description: Incremental (i.e., baseline-corrected) mean area under the 24-hour plasma glucagon concentration curve with a pre-test, non-fasting plasma glucagon value as baseline. (Sample times: 0, 30 min, 2 hours [dinner], 2 hours 45 min, 3 hours, 4 hours, 9 hours, 12 hours, 14 hours, 16 hours [breakfast], 16 hours 45 min, 17 hours, 18 hours, 20 hours [lunch], 20 hours 45 min, 21 hours, 23 hours, 24 hours).
Time Frame: 24 h
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: pmol/L*h
Arm/Group | Placebo & Regular Insulin | Pramlintide & Regular Insulin
Number analyzed (Participants) | 26 | 26
pmol/L*h | -14.954 (58.9024) | -16.055 (69.2684)

11. Secondary Outcome: Fasting Plasma Glucose Concentration
Description: Fasting plasma glucose concentration at 0600 hours (6:00 AM)
Time Frame: 12 hours after dinner meal
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Placebo & Regular Insulin | Pramlintide & Regular Insulin
Number analyzed (Participants) | 26 | 26
mmol/L | 7.794 [6.631 to 9.162] | 8.459 [7.196 to 9.943]
Statistical Analysis 1: Comparison: Placebo & Regular Insulin vs Pramlintide & Regular Insulin; Test type: Superiority or Other; p = 0.3730, Linear mixed effects model; LS mean ratio (pramlintide/placebo) = 1.085, 95% CI 2-sided [0.901 to 1.307]

12. Secondary Outcome: Pharmacokinetics of Insulin as Demonstrated by 24-hour Plasma Insulin Area Under the Plasma Concentration-time Curve (AUC)
Description: Mean areas under the plasma insulin concentration curves for the 24-hour periods of pramlintide and placebo administration (Sample times: -15 min, 0, 30 min, 1 hour 30 min, 2 hours [dinner], 2 hours 15 min, 2 hours 30 min, 2 hours 45 min, 3 hours, 4 hours, 5 hours, 6 hours, 9 hours, 12 hours, 15 hours, 16 hours [breakfast], 16 hours 15 min, 16 hours 30 min, 16 hours 45 min, 17 hours, 18 hours, 19 hours, 20 hours [lunch], 24 hours).
Time Frame: 24 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mU/L*h
Arm/Group | Placebo & Regular Insulin | Pramlintide & Regular Insulin
Number analyzed (Participants) | 26 | 26
mU/L*h | 380.525 (178.2360) | 377.324 (176.7569)

13. Secondary Outcome: Pharmacokinetics of Insulin as Demonstrated by 24-hour Average Plasma Insulin Concentration.
Description: Mean values of the average plasma insulin concentrations over the 24-hour periods of pramlintide and placebo administration. (Sample times: -15 min, 0, 30 min, 1 hour 30 min, 2 hours [dinner], 2 hours 15 min, 2 hours 30 min, 2 hours 45 min, 3 hours, 4 hours, 5 hours, 6 hours, 9 hours, 12 hours, 15 hours, 16 hours [breakfast], 16 hours 15 min, 16 hours 30 min, 16 hours 45 min, 17 hours, 18 hours, 19 hours, 20 hours [lunch], 24 hours).
Time Frame: 24 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | Placebo & Regular Insulin | Pramlintide & Regular Insulin
Number analyzed (Participants) | 26 | 26
mIU/L | 15.855 (7.4265) | 15.722 (7.3649)

14. Secondary Outcome: Pharmacokinetics of Insulin as Demonstrated by Maximum Plasma Insulin Concentration
Description: Mean maximum plasma insulin concentrations over the 24-hour periods of pramlintide and placebo administration. (Sample times: -15 min, 0, 30 min, 1 hour 30 min, 2 hours [dinner], 2 hours 15 min, 2 hours 30 min, 2 hours 45 min, 3 hours, 4 hours, 5 hours, 6 hours, 9 hours, 12 hours, 15 hours, 16 hours [breakfast], 16 hours 15 min, 16 hours 30 min, 16 hours 45 min, 17 hours, 18 hours, 19 hours, 20 hours [lunch], 24 hours).
Time Frame: 24 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mIU/L
Arm/Group | Placebo & Regular Insulin | Pramlintide & Regular Insulin
Number analyzed (Participants) | 26 | 26
mIU/L | 33.144 (17.0950) | 32.838 (16.2315)

15. Secondary Outcome: Pharmacokinetics of Insulin as Demonstrated by the Time to the Maximum Plasma Insulin Concentration
Description: Mean time to maximum plasma insulin concentrations over the 24-hour periods of pramlintide and placebo administration. (Sample times: -15 min, 0, 30 min, 1 hour 30 min, 2 hours [dinner], 2 hours 15 min, 2 hours 30 min, 2 hours 45 min, 3 hours, 4 hours, 5 hours, 6 hours, 9 hours, 12 hours, 15 hours, 16 hours [breakfast], 16 hours 15 min, 16 hours 30 min, 16 hours 45 min, 17 hours, 18 hours, 19 hours, 20 hours [lunch], 24 hours).
Time Frame: 24 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: h
Arm/Group | Placebo & Regular Insulin | Pramlintide & Regular Insulin
Number analyzed (Participants) | 26 | 26
h | 10.556 (7.3466) | 11.653 (7.6175)

ADVERSE EVENTS:
Time Frame: Over two 24-hour treatment periods with a 2-week washout period between periods.
Description: This was a crossover study.
Arm/Group | Placebo & Regular Insulin | Pramlintide & Regular Insulin
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/32
Other Adverse Events (participants affected / at risk) | 9/28 | 22/32
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo & Regular Insulin (N=28) | Pramlintide & Regular Insulin (N=32)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 6 (6)
Nausea (Gastrointestinal disorders) | 2 (2) | 14 (14)
Cardiovascular disorder (Cardiac disorders) | 0 (0) | 1 (1)
Vitreous Detachment (Eye disorders) | 1 (1) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Tremor (Nervous system disorders) | 2 (3) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 8 (9)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pruritus allergic (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Scab (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Due to the unavailability of the pramlintide assay, no data are presented for pramlintide PK parameters, and changes in pramlintide concentration could not be related to changes in insulin, plasma glucose, glucagon, or triglycerides.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No